CLINICAL TRIAL: NCT02623257
Title: A Diagnostic Study to Determine the Prevalence of Epidermal Growth Factor Receptor Mutations Assessed With Circulating Tumor DNA Samples in Advanced Non-small Cell Lung Cancer
Brief Title: EGFR Mutations on ctDNA in Patients With Advanced NSCLC
Status: Completed | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 20154701
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer Stage III; Non-Small-Cell Lung Cancer Metastatic
Keywords: Non-small Cell Lung Cancer; circulating tumor DNA; amplification refractory mutation system
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: mutation detection
Other: ARMS
Genetic: ctDNA analysis

SUMMARY:
The study aims to explore the prevalence of EGFR mutations assessed with ctDNA samples in advanced NSCLC, who had received ≤ 1 prior systemic chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIB/IV NSCLC;
* Patient had received ≤ 1 prior systemic chemotherapy regimens;
* Provision of blood (plasma) sample for ctDNA testing;
* Patient must be able to comply with the protocol;

Exclusion Criteria:

* Prior received ≥2 systemic chemotherapy regimens;
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease);
* Histologically confirmed small cell lung cancer or other metastatic tumors;
* Patient with no histologic or cytological diagnosis;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 1055 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with EGFR mutation detected by amplification refractory mutation system (ARMS) assay | up to 2 years
  The investigators will describe the proportion of EGFR mutation on ctDNA detected by ARMS assay in patients with non-small cell lung cancer (NSCLC)

SECONDARY OUTCOMES:
Distribution of EGFR mutation by ARMS assays among the different Clinical characteristics | up to 2 years
  The investigators will employ chi-square test to analyze the distribution of EGFR mutation by ARMS in NSCLC patients among the different characteristics including smoking status, gender, age, PS score, and tumor stage
Proportion of treatment-naive patients with EGFR mutation detected by amplification refractory mutation system (ARMS) assay | up to 2 years
  The investigators will describe the proportion of EGFR mutation on ctDNA detected by ARMS assay in treatment-naive patients with non-small cell lung cancer (NSCLC)
Proportion of patients after first-line chemotherapy failure with EGFR mutation detected by amplification refractory mutation system (ARMS) assay | up to 2 years
  The investigators will describe the proportion of EGFR mutation on ctDNA detected by ARMS assay in non-small cell lung cancer (NSCLC) patients after first-line chemotherapy failure

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China